CLINICAL TRIAL: NCT00077376
Title: A Phase II Trial of Trastuzumab Plus Weekly Ixabepilone(BMS-247550) and Carboplatin in Patients With HER2/Neu-Positive Metastatic Breast Cancer
Brief Title: Trastuzumab, Ixabepilone, and Carboplatin in Treating Patients With HER2/Neu-Positive Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02946; NCI-2012-02946 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); U10CA023318 (NIH); E2103 (Other: Eastern Cooperative Oncology Group); E2103 (Other: CTEP); U10CA021115 (NIH)
Record Dates: First submitted 2004-02-10; First posted 2004-02-12 (Estimated); Results first posted 2011-04-04 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2012-12

CONDITIONS: HER2-positive Breast Cancer; Male Breast Cancer; Recurrent Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms | interventions — Trastuzumab; ixabepilone; Carboplatin

ARMS (1):
- Treatment (trastuzumab, ixabepilone, carboplatin) (Experimental): Induction therapy: Patients receive trastuzumab (Herceptin®) IV over 30 minutes* on days 1, 8, 15, and 22 and ixabepilone IV over 1 hour and carboplatin IV over 1 hour on days 1, 8, and 15. Treatment repeats every 28 days for up to 6 courses in the absence of unacceptable toxicity.
  NOTE: *Trastuzumab is given over 90 minutes on day 1 of course 1 (induction therapy) only.
  Maintenance therapy: Patients receive trastuzumab IV over 90 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: trastuzumab; Drug: ixabepilone; Drug: carboplatin; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: trastuzumab — Given IV
  Other Names: anti-c-erB-2; Herceptin; MOAB HER2
Drug: ixabepilone — Given IV
  Other Names: BMS-247550; epothilone B lactam; Ixempra
Drug: carboplatin — Given IV
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well giving trastuzumab together with ixabepilone and carboplatin works in treating patients with HER2/neu-positive metastatic breast cancer. Monoclonal antibodies, such as trastuzumab, can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Drugs used in chemotherapy, such as ixabepilone and carboplatin, work in different ways to stop tumor cells from dividing so they stop growing or die. Combining trastuzumab with ixabepilone and carboplatin may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the response rate (as determined by RECIST criteria) to combination therapy with Ixabepilone (BMS-247550), trastuzumab, and carboplatin in patients with metastatic breast cancer known to overexpress HER2.

SECONDARY OBJECTIVES:

I. To determine time to disease progression (TTP) and time to treatment failure (TTF) after treatment with Ixabepilone (BMS-247550), trastuzumab and carboplatin in patients with metastatic breast cancer known to overexpress HER2.

II. To determine the toxicity of combination therapy with Ixabepilone (BMS-247550), trastuzumab and carboplatin in patients with metastatic breast cancer known to overexpress HER2.

III. To evaluate overall survival (OS) of combination therapy with Ixabepilone (BMS-247550), trastuzumab, and carboplatin in patients with metastatic breast cancer known to overexpress HER2.

IV. To correlate levels of phospho-STAT3 with levels of HER2, Survivin and EGFR expression as measured in tissue by immunohistochemistry.

OUTLINE: This is a multicenter study.

Induction therapy: Patients receive trastuzumab (Herceptin®) IV over 30 minutes* on days 1, 8, 15, and 22 and ixabepilone IV over 1 hour and carboplatin IV over 1 hour on days 1, 8, and 15. Treatment repeats every 28 days for up to 6 courses in the absence of unacceptable toxicity.

NOTE: *Trastuzumab is given over 90 minutes on day 1 of course 1 (induction therapy) only.

Maintenance therapy: Patients receive trastuzumab IV over 90 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years and then every 6 months for 3 years from study entry.

PROJECTED ACCRUAL: A total of 10-60 patients will be accrued for this study within 1-6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed adenocarcinoma of the breast which is metastatic and is known to overexpress HER2/neu who have received no prior chemotherapy for metastatic breast cancer; prior hormonal therapy for metastatic disease is allowed; NOTE: for this protocol, HER2 overexpression will be defined as 3+ HER2 positivity as measured by immunohistochemistry using the HercepTest (DAKO) or HER2 gene amplification as measured by fluorescent in-situ hybridization (FISH, e.g. Vysis); representative diagnostic tissue must be submitted for central diagnostic review
* Patients must not be pregnant or breast feeding because of the teratogenic potential of these drugs; it is recommended that all females of childbearing potential have a blood test or urine study within 2 weeks prior to registration to rule out pregnancy; women of childbearing potential and sexually active males must be strongly advised to use an accepted and effective non-hormonal method of contraception
* Patients must have at least one objective measurable disease parameter; baseline measurements and evaluations using RECIST criteria guidelines must be obtained within 4 weeks prior to registration to the study; NOTE: all areas of disease should be recorded and followed
* Patients must have an ECOG performance status of 0 or 1
* Patients must be disease free of prior malignancy for >= 5 years with the exception of curatively treated basal cell carcinoma or squamous cell carcinomas of the skin or carcinoma in situ of the cervix
* Patients must not have a history of untreated brain metastasis or brain metastasis currently undergoing radiation; patients with brain metastasis representing the sole site of disease are not eligible for this study; patients with previously treated brain metastasis who have responded to brain radiotherapy and/or surgery and continue in response are eligible provided the brain is not the only site of measurable disease
* Patients must not have peripheral neuropathy of any grade
* Patients must not have a history of prior severe (grade 3 or 4) hypersensitivity reaction to a drug formulated in polyoxyethylated castor oil (Cremophor EL)
* Patients must have left ventricular ejection fraction by MUGA scan or echocardiogram that is at or above the lower institutional limits of normal obtained within 6 weeks prior to registration
* Patients must not have a history of New York Heart Association class 3 or 4 heart failure
* Serum creatinine =< 1.5 mg/dl
* Granulocytes >= 1500/mm^3
* Platelets >= 100,000/mm^3
* SGOT(AST) and SGPT(ALT) =< 1.5 x upper limit of normal (unless liver is involved by tumor, in which case SGOT(AST) and SGPT(ALT) can be =< 2.0 x upper limit of normal)
* Patients must have no history of prior therapy with trastuzumab (Herceptin), Ixabepilone (BMS-247550) or carboplatin for metastatic disease; patients who develop metastatic disease =< 6 months after completing adjuvant trastuzumab (Herceptin), paclitaxel, docetaxel, carboplatin, or Ixabepilone (BMS-247550) are considered to have had prior therapy for metastatic disease and are excluded from study participation
* Patients must not have received a cumulative dose of doxorubicin of greater than 360 mg/m^2 or epirubicin of greater than 640 mg/m^2
* Concurrent use of hormonal therapy is not permitted; concurrent radiation therapy is not permitted; hormonal therapy must have been discontinued >= 1 week prior to registration; radiation therapy must have been completed >= 2 weeks prior to registration
* Patients may have had prior radiation therapy, but the previously irradiated tumors cannot be used to assess a clinical response; patients will not be eligible if they do not have other areas of measurable disease; an exception will be given for patients who have had tumor recurrence in an area that received adjuvant radiation treatments, such as the axilla or chest wall

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2005-03; Primary Completion 2009-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stacy Moulder, Principal Investigator — Eastern Cooperative Oncology Group
Locations (1):
- Eastern Cooperative Oncology Group, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on March 19th, 2004. Accrual was suspended on December 16th, 2004 after reaching the first stage accrual goal. After a pre-planned toxicity analysis, accrual resumed on March 4th, 2005. The study was completed on March 24th, 2006, after accruing 61 patients.
Groups:
- Trastuzumab/Ixabepilone/Carboplatin: During the induction phase, patients were treated with Ixabepilone (BMS-247550) 15mg/m2 intravenously (IV) followed by carboplatin (AUC=2 IV) on days 1, 8 and 15 of a 28-day cycle for a maximum of 6 cycles. Trastuzumab was administered weekly (4mg/kg loading dose then 2mg/kg IV) starting on day 1. Routine premedication included H1 blocker (diphenhydramine 50 mg orally (PO) or IV), H2 blocker (ranitidine 150 mg PO or 50 mg IV or another equivalent H2 blocker), and at least a 5-HT3 antagonist and dexamethasone.
  After completion of 24 weekly trastuzumab doses (induction therapy), trastuzumab were given at a dose of 6 mg/kg IV every 3 weeks (maintenance therapy) beginning one week after the 24th weekly dose. Trastuzumab were repeated every 21 days until disease progression or prohibitive toxicity.
Period: Overall Study
Arm/Group | Trastuzumab/Ixabepilone/Carboplatin
Started | 61
Treated | 59
HER2+ in Central Testing | 39
Completed | 39
Not Completed | 22
Not completed — Adverse Event | 8
Not completed — Withdrawal by Subject | 2
Not completed — Death | 1
Not completed — Physician Decision | 1
Not completed — Alternative therapy | 5
Not completed — Complicating disease | 1
Not completed — Still on treatment | 1
Not completed — Symptomatic deterioration | 1
Not completed — Surgery | 1
Not completed — Insurance ran out | 1

BASELINE CHARACTERISTICS:
Arm/Group | Trastuzumab/Ixabepilone/Carboplatin
Number analyzed (Participants) | 59
Age, Continuous [Median (Full Range); unit: years] — All treated patients
  years | 51 [24 to 81]
Age, Continuous [Median (Full Range); unit: years] — HER2+ patients only
  years | 54 [24 to 81]
Sex: Female, Male [Count of Participants; unit: Participants] — All treated patients
  Participants
    Female | 59
    Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response for HER2+ Patients (Best Objective Response a Patient Has Ever Experienced on Study)
Description: To assess objective response, it is necessary to estimate the overall tumor burden at baseline to which subsequent measurements will be compared. The same method of assessment and the same technique should be used to characterize each lesion at baseline and during follow-up.
  The best overall response based on RECIST is the best response recorded from registration until disease progression/recurrence, taking as reference for progressive disease the smallest measurements recorded since registration. The best response was determined based on the tumor responses in target and nontarget lesions, with or without new lesions. To be assigned a status of complete or partial response, changes in tumor measurements must be confirmed by repeat assessments performed no less than 4 weeks after the criteria for response are first met. To be assigned a status of stable disease, measurements must have met the stable disease criteria at least once after study entry at a minimum interval of 8 weeks.
Time Frame: Assessed every 3 cycles during induction therapy and every 6 cycles during maintenance therapy until disease progression or up to 5 years
Population: HER2+ patients
Measure: Number; unit: Participants
Arm/Group | Trastuzumab/Ixabepilone/Carboplatin
Number analyzed (Participants) | 39
Participants
  Complete Response | 3
  Partial Response | 13
  No Change/ Stable | 10
  Progression | 11
  Unevaluable | 2
Statistical Analysis 1: Comparison: Trastuzumab/Ixabepilone/Carboplatin; Test type: Superiority or Other; Objective response rate = 41, 95% CI 2-sided [26 to 58]

2. Secondary Outcome: Objective Response for All Treated Patients (the Best Response a Patient Has Ever Experienced on Study)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: All treated patients
Measure: Number; unit: Participants
Arm/Group | Trastuzumab/Ixabepilone/Carboplatin
Number analyzed (Participants) | 59
Participants
  Compelete Response | 4
  Partial Response | 22
  No Change/ Stable | 15
  Progression | 16
  Unevaluable | 2
Statistical Analysis 1: Comparison: Trastuzumab/Ixabepilone/Carboplatin; Test type: Superiority or Other; Objective response rate = 44, 95% CI 2-sided [31 to 58]

3. Secondary Outcome: Time to Disease Progression for HER2+ Patients
Description: This interval will be measured from the date of entry on the study to the appearance of new metastatic lesions or objective tumor progression based on RECIST. Patients progression-free at last follow-up were censored.
Time Frame: as for outcome 1
Population: HER2+ patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trastuzumab/Ixabepilone/Carboplatin
Number analyzed (Participants) | 39
Months | 7.1 [5.5 to 9.7]

4. Secondary Outcome: Time to Disease Progression for All Treated Patients
Description: as for outcome 3
Time Frame: as for outcome 1
Population: All treated patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trastuzumab/Ixabepilone/Carboplatin
Number analyzed (Participants) | 59
Months | 8.2 [6.3 to 9.9]

5. Secondary Outcome: Time to Treatment Failure for HER2+ Patients
Description: Time from study entry to the date at which a patient was removed from treatment due to progression, toxicity, refusal or death. If a patient was considered to be a major treatment violation or was taken off study as a non-protocol failure, the patient would be censored on the date he/she was removed from treatment.
Time Frame: Assessed every cycle until treatment discontinuation
Population: HER2+ patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trastuzumab/Ixabepilone/Carboplatin
Number analyzed (Participants) | 39
Months | 5.4 [5.3 to 6.2]

6. Secondary Outcome: Time to Treatment Failure for All Treated Patients
Description: as for outcome 5
Time Frame: Assessed every cycle until treatment discontinuation
Population: All treated patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trastuzumab/Ixabepilone/Carboplatin
Number analyzed (Participants) | 59
Months | 5.9 [5.3 to 7.6]

7. Secondary Outcome: Kaplan-Meier Estimate of Overall Survival at 3 Years for HER2+ Patients
Description: Survival estimate from the Kaplan-Meier curve of the proportion of patients alive at 3 years.
Time Frame: Assessed every 3 months for 2 years, then every 6 months for 3 years
Population: HER2+ patients
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Trastuzumab/Ixabepilone/Carboplatin
Number analyzed (Participants) | 39
Percentage of Participants | 50 [33.3 to 66.0]

8. Secondary Outcome: Kaplan-Meier Estimate of Overall Survival at 3 Years for All Treated Patients
Description: Survival estimate from the Kaplan-Meier curve of the proportion of patients alive at 3 years.
Time Frame: Assessed every 3 months for 2 years, then every 6 months for 3 years
Population: All treated patients
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Trastuzumab/Ixabepilone/Carboplatin
Number analyzed (Participants) | 59
Percentage of Participants | 48 [34.2 to 61.6]

ADVERSE EVENTS:
Time Frame: Assessed every cycle (1 induction cycle = 4 weeks, 1 maintenance cycle = 3 weeks) while on treatment and for 30 days after the end of treatment.
Arm/Group | Trastuzumab/Ixabepilone/Carboplatin
Serious Adverse Events (participants affected / at risk) | 39/59
Other Adverse Events (participants affected / at risk) | 59/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab/Ixabepilone/Carboplatin (N=59)
Allergic reaction (Immune system disorders) | 2
Anemia (Blood and lymphatic system disorders) | 7
Leukopenia (Investigations) | 19
Neutropenia (Investigations) | 29
Thrombocytopenia (Investigations) | 8
Hematologic-other (Blood and lymphatic system disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Fatigue (General disorders) | 7
Weight loss (Investigations) | 1
Death NOS (General disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 3
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 2
Infection with Grade 0-2 neutrophils, urinary tract (Infections and infestations) | 2
Alkaline phosphatase increased (Investigations) | 1
AST increased (Investigations) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Neuropathy-sensory (Nervous system disorders) | 4
Syncope (Nervous system disorders) | 1
Abdomen, pain (Gastrointestinal disorders) | 1
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 1
Joint, pain (Musculoskeletal and connective tissue disorders) | 1
Muscle, pain (Musculoskeletal and connective tissue disorders) | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab/Ixabepilone/Carboplatin (N=59)
Allergic reaction (Immune system disorders) | 8
Anemia (Blood and lymphatic system disorders) | 55
Leukopenia (Investigations) | 54
Neutropenia (Investigations) | 44
Thrombocytopenia (Investigations) | 37
Left ventricular systolic dysfunction (Cardiac disorders) | 6
Fatigue (General disorders) | 51
Fever w/o neutropenia (General disorders) | 5
Insomnia (Psychiatric disorders) | 7
Rigors/chills (General disorders) | 3
Sweating (Skin and subcutaneous tissue disorders) | 3
Weight loss (Investigations) | 10
Dry skin (Skin and subcutaneous tissue disorders) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 33
Pruritus/itching (Skin and subcutaneous tissue disorders) | 4
Rash/desquamation (Skin and subcutaneous tissue disorders) | 10
Hot flashes (Vascular disorders) | 3
Anorexia (Metabolism and nutrition disorders) | 22
Constipation (Gastrointestinal disorders) | 24
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 33
Dyspepsia (Gastrointestinal disorders) | 11
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 17
Nausea (Gastrointestinal disorders) | 42
Taste disturbance (Nervous system disorders) | 21
Vomiting (Gastrointestinal disorders) | 20
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 5
Infection with Grade 0-2 neutrophils, skin (Infections and infestations) | 3
Infection with Grade 0-2 neutrophils, urinary tract (Infections and infestations) | 3
Edema limb (General disorders) | 10
Hypoalbuminemia (Metabolism and nutrition disorders) | 3
Alkaline phosphatase increased (Investigations) | 17
ALT increased (Investigations) | 24
AST increased (Investigations) | 20
Bilirubin increased (Investigations) | 4
Creatinine increased (Investigations) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 28
Hypoglycemia (Metabolism and nutrition disorders) | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 4
Dizziness (Nervous system disorders) | 7
Anxiety (Psychiatric disorders) | 3
Neuropathy-motor (Nervous system disorders) | 4
Neuropathy-sensory (Nervous system disorders) | 36
Abdomen, pain (Gastrointestinal disorders) | 6
Back, pain (Musculoskeletal and connective tissue disorders) | 3
Chest/thoracic pain NOS (General disorders) | 5
Head/headache (Nervous system disorders) | 8
Joint, pain (Musculoskeletal and connective tissue disorders) | 14
Muscle, pain (Musculoskeletal and connective tissue disorders) | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less